CLINICAL TRIAL: NCT05286333
Title: Identification of Risk Factors for Recurrence of Low Back Pain and Occupational Repercussions Among Beneficiaries of a Multidisciplinary Follow-up Shared Between Physical and Rehabilitation Medicine and Occupational Medicine: a Monocentric Prospective Study
Brief Title: Identification of Risk Factors for Recurrence of Low Back Pain and Occupational Repercussions
Acronym: LORET
Status: Recruiting | Type: Observational
Sponsor: Fondation Ildys (Other)
Collaborators: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: ID-RCB 2021-A02371-40
Record Dates: First submitted 2022-02-25; First posted 2022-03-18 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Low back pain (LBP) is the leading cause of disability and one of the most common reasons for physician visits in primary care, with a 33 % rate of recurrence during the first year, converting LBP into a chronic condition.

The french High healthy authority recommend early occupational oriented intervention associated with a multidisciplinary rehabilitation program.

However even if these recommendations are taken into appropriate account, risk for recurrence of Low back pain and occupational repercussions often occured.

This study aims to identify the risk factor(s) of sick leave after a rehabilitation stay in outpatients and thus adapt cares provided to the patients in respect of their needs and expectations.

ELIGIBILITY:
Inclusion Criteria:

* men and women over 18 years old
* able to understand and respect the protocol requirement
* who signed the consent prior to any other procedure protocol
* patients suffering from chronic lower back or lumbo-radicular pain since more than 3 months
* employee bellow 3 years before retirement
* patients included in a multidisciplinary rehabilitation program and occupational medicine

Exclusion Criteria:

* major patients under guardianship/curator/legal protection
* pregnant patients
* obese patients with BMI (body mass index) > 35 (grade 2)
* patients suffering from neurological pathology
* patients suffering from chronic lower back or lumbo-radicular pain since less than 3 months
* patients suffering from chronic lower back pain with inflammatory or tumoral or infectious ethiology

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All the beneficiaries of the multidisciplinary follow-up shared between the physical and rehabilitation medicine and occupational medicine, will be elligible in this study.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Recurrence of sick leaves induced by lower back pain | 3 months after the rehabilitation program
  Number of sick leaves induced by lower back pain after the rehabilitation program
Recurrence of sick leaves induced by lower back pain | 6 months after the rehabilitation program
  Number of sick leaves induced by lower back pain after the rehabilitation program
Recurrence of sick leaves induced by lower back pain | 9 months after the rehabilitation program
  Number of sick leaves induced by lower back pain after the rehabilitation program
Recurrence of sick leaves induced by lower back pain | 12 months after the rehabilitation program
  Number of sick leaves induced by lower back pain after the rehabilitation program

SECONDARY OUTCOMES:
Risk factor analysis of recurrence of sick leaves induced by lower back pain (1) | Baseline
  demography (sexe and age) will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (2) | Baseline
  anthropometric data (weight, BMI) will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (3) | Baseline
  quality of life,evaluated by Oswestry scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (3) | 3 months after the rehabilitation program
  quality of life,evaluated by Oswestry scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (3) | 6 months after the rehabilitation program
  quality of life,evaluated by Oswestry scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (3) | 9 months after the rehabilitation program
  quality of life,evaluated by Oswestry scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (3) | 12 months after the rehabilitation program
  quality of life,evaluated by Oswestry scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (4) | Baseline
  Physiological state, evaluated by hospital anxiety and depression scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (4) | 3 months after the rehabilitation program
  Physiological state, evaluated by hospital anxiety and depression scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (4) | 6 months after the rehabilitation program
  Physiological state, evaluated by hospital anxiety and depression scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (4) | 9 months after the rehabilitation program
  Physiological state, evaluated by hospital anxiety and depression scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (4) | 12 months after the rehabilitation program
  Physiological state, evaluated by hospital anxiety and depression scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (5) | Baseline
  physical activity, evaluated by Ricci & gagnon questionnaire, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (5) | 3 months after the rehabilitation program
  physical activity, evaluated by Ricci & gagnon questionnaire, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (5) | 6 months after the rehabilitation program
  physical activity, evaluated by Ricci & gagnon questionnaire, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (5) | 9 months after the rehabilitation program
  physical activity, evaluated by Ricci & gagnon questionnaire, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (5) | 12 months after the rehabilitation program
  physical activity, evaluated by Ricci & gagnon questionnaire, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (6) | Baseline
  Pain, evaluated with a visual analog scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (6) | 3 months after the rehabilitation program
  Pain, evaluated with a visual analog scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (6) | 6 months after the rehabilitation program
  Pain, evaluated with a visual analog scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (6) | 9 months after the rehabilitation program
  Pain, evaluated with a visual analog scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (6) | 12 months after the rehabilitation program
  Pain, evaluated with a visual analog scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (7) | Baseline
  Impact of lower back pain on wellbeing, evaluated with Dallas questionnaire, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (7) | 3 months after the rehabilitation program
  Impact of lower back pain on wellbeing, evaluated with Dallas questionnaire, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (7) | 6 months after the rehabilitation program
  Impact of lower back pain on wellbeing, evaluated with Dallas questionnaire, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (7) | 9 months after the rehabilitation program
  Impact of lower back pain on wellbeing, evaluated with Dallas questionnaire, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (7) | 12 months after the rehabilitation program
  Impact of lower back pain on wellbeing, evaluated with Dallas questionnaire, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (8) | Baseline
  stress at work, evaluated with Karasek scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (8) | 3 months after the rehabilitation program
  stress at work, evaluated with Karasek scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (8) | 6 months after the rehabilitation program
  stress at work, evaluated with Karasek scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (8) | 9 months after the rehabilitation program
  stress at work, evaluated with Karasek scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (8) | 12 months after the rehabilitation program
  stress at work, evaluated with Karasek scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (9) | Baseline
  Fear and beliefs, evaluated with FABQ (Fear-avoidance beliefs questionnaire) scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (9) | 3 months after the rehabilitation program
  Fear and beliefs, evaluated with FABQ (Fear-avoidance beliefs questionnaire) scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (9) | 6 months after the rehabilitation program
  Fear and beliefs, evaluated with FABQ (Fear-avoidance beliefs questionnaire) scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (9) | 9 months after the rehabilitation program
  Fear and beliefs, evaluated with FABQ (Fear-avoidance beliefs questionnaire) scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (9) | 12 months after the rehabilitation program
  Fear and beliefs, evaluated with FABQ (Fear-avoidance beliefs questionnaire) scale, will be analysed as risk factor of recurrence
Risk factor analysis of recurrence of sick leaves induced by lower back pain (10) | Baseline
  locomotor capacity (flexibility and endurance) will be analysed as risk factor of recurrence.
Risk factor analysis of recurrence of sick leaves induced by lower back pain (10) | 6 months after the rehabilitation program
  locomotor capacity (flexibility and endurance) will be analysed as risk factor of recurrence.
Risk factor analysis of recurrence of sick leaves induced by lower back pain (10) | 12 months after the rehabilitation program
  locomotor capacity (flexibility and endurance) will be analysed as risk factor of recurrence.
Risk factor analysis of recurrence of sick leaves induced by lower back pain (11) | Baseline
  neurological impact (tendon reflex) will be analysed as risk factor of recurrence.
Risk factor analysis of recurrence of sick leaves induced by lower back pain (11) | 6 months after the rehabilitation program
  neurological impact (tendon reflex) will be analysed as risk factor of recurrence.
Risk factor analysis of recurrence of sick leaves induced by lower back pain (11) | 12 months after the rehabilitation program
  neurological impact (tendon reflex) will be analysed as risk factor of recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Bourseul, MD, Principal Investigator — Fondation Ildys
Locations (1):
- Centre de Perharidy, Roscoff, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palazzo C, Ravaud JF, Papelard A, Ravaud P, Poiraudeau S. The burden of musculoskeletal conditions. PLoS One. 2014 Mar 4;9(3):e90633. doi: 10.1371/journal.pone.0090633. eCollection 2014. PMID 24595187
- [Background] Cougot B, Petit A, Paget C, Roedlich C, Fleury-Bahi G, Fouquet M, Menu P, Dubois C, Geraut C, Roquelaure Y, Tripodi D. Chronic low back pain among French healthcare workers and prognostic factors of return to work (RTW): a non-randomized controlled trial. J Occup Med Toxicol. 2015 Oct 29;10:40. doi: 10.1186/s12995-015-0082-5. eCollection 2015. PMID 26516339
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Lawlis GF, Cuencas R, Selby D, McCoy CE. The development of the Dallas Pain Questionnaire. An assessment of the impact of spinal pain on behavior. Spine (Phila Pa 1976). 1989 May;14(5):511-6. doi: 10.1097/00007632-198905000-00007. PMID 2524890
- [Background] da Silva T, Mills K, Brown BT, Pocovi N, de Campos T, Maher C, Hancock MJ. Recurrence of low back pain is common: a prospective inception cohort study. J Physiother. 2019 Jul;65(3):159-165. doi: 10.1016/j.jphys.2019.04.010. Epub 2019 Jun 14. PMID 31208917
- [Background] da Silva T, Mills K, Brown BT, Herbert RD, Maher CG, Hancock MJ. Risk of Recurrence of Low Back Pain: A Systematic Review. J Orthop Sports Phys Ther. 2017 May;47(5):305-313. doi: 10.2519/jospt.2017.7415. Epub 2017 Mar 29. PMID 28355981
- [Background] Yvanes-Thomas M, Calmels P, Bethoux F, Richard A, Nayme P, Payre D, Laurent B. Validity of the French-language version of the Quebec back pain disability scale in low back pain patients in France. Joint Bone Spine. 2002 Jun;69(4):397-405. doi: 10.1016/s1297-319x(02)00415-3. PMID 12184438
- [Background] Karasek RA, Theorell T, Schwartz JE, Schnall PL, Pieper CF, Michela JL. Job characteristics in relation to the prevalence of myocardial infarction in the US Health Examination Survey (HES) and the Health and Nutrition Examination Survey (HANES). Am J Public Health. 1988 Aug;78(8):910-8. doi: 10.2105/ajph.78.8.910. PMID 3389427
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Background] Chaory K, Fayad F, Rannou F, Lefevre-Colau MM, Fermanian J, Revel M, Poiraudeau S. Validation of the French version of the fear avoidance belief questionnaire. Spine (Phila Pa 1976). 2004 Apr 15;29(8):908-13. doi: 10.1097/00007632-200404150-00018. PMID 15082995